CLINICAL TRIAL: NCT00222326
Title: The Effect of a Physiotherapy Treatment Program on Pelvic Function Following Gynaecological Surgery
Brief Title: The Effect of Physiotherapy Treatment Following Gynaecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Mary Galea, Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-15-10-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Vaginal Hysterectomy; Pelvic Organ Prolapse Vaginal Surgery
Keywords: Hysterectomy; Prolapse; Pelvic floor muscles; Bladder; Bowel
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor muscle training (Experimental): Pelvic floor muscle training: clinic and rooms exercise training
  Interventions: Behavioral: Pelvic floor muscle training and lifestyle modification
- Usual care (No Intervention): Usual care as provided by the surgeon and hospital staff

INTERVENTIONS:
Behavioral: Pelvic floor muscle training and lifestyle modification
  Arms: Pelvic floor muscle training

SUMMARY:
Optimal pelvic floor muscle function is known to assist bladder and bowel function and control, pelvic organ support, as well as other areas of health. It is also known that problems in some of tehse areas can be a consequence of pelvic surgery. By addressing the requirements for good bladder and bowel function/control, and organ support in the early post-surgery phase when tissue repair and scar formation are critical, it is proposed that there will be a rduction in the longterm prevalence of bladder problems, bowel difficulties and weakened pelvic floor and abdominal muscles in post-surgery patients. This study is a randomised controlled trial to compare patients undergoing a physiotherapy-supervised pelvic floor muscle training and behavioural therapy program with a control group. It is hypothesised that at the 12 month post-operative follow-up assessment, the treatment group will demonstrate better outcomes in bladder and bowel function and control, as well as stronger pelvic floor muscle contractile strength than the control group.

DETAILED DESCRIPTION:
Optimal pelvic floor muscle function is known to assist bladder and bowel function and control, pelvic organ support, as well as other areas of pelvic health. It is also known that problems in some of these areas can develop after pelvic surgery. By addressing the requirements for good bladder and bowel function/control, and organ support in the early post-surgical phase when tissue repair and scar formation are critical, it is proposed that there will be a reduction in the long-term prevalence of bladder and bowel dysfunction, and weak pelvic floor and abdominal muscles in post-surgical patients. There have been no previous studies investigating whether a physiotherapy intervention can assist pelvic function in this group of surgical patients.

This study aims to investigate the effect of a physiotherapy treatment program on pelvic function following gynaecological surgery.

Comparisons: Pre- and post-operative physiotherapy treatment vs no treatment following gynaecological surgery.

Outcome measures: Pelvic floor muscle strength, urine leakage, quality of life, sexual functioning, general fitness, measured at 3, 6 and 12 months post-operatively

ELIGIBILITY:
Inclusion Criteria:

* undergoing vaginal gynaecological surgery, for hysterectomy or prolapse repair

Exclusion Criteria:

* surgery for malignancy
* anti-incontinence surgery
* laparotomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-07; Primary Completion 2006-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Bladder symptom (prevalence and bother) questionnaire. | Pre-operative compared to 12 months post-operative
  A questionnaire about bladder symptoms
Prolapse symptom (prevalence and bother) questionnaire. | Pre-operative compared to 12 months post-operative
  A questionnaire about prolapse symptoms

SECONDARY OUTCOMES:
Pelvic floor muscle strength. | Pre-operative compared to 12 months post-operative
  Strength assessed via digital muscle testing

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Galea, PhD, Principal Investigator — The University of Melbourne, Australia
Locations (1):
- School of Physiotherapy, The University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Frawley HC, Galea MP, Phillips BA. Survey of clinical practice: pre- and postoperative physiotherapy for pelvic surgery. Acta Obstet Gynecol Scand. 2005 May;84(5):412-8. doi: 10.1111/j.0001-6349.2005.00776.x. PMID 15842203
- [Result] Frawley HC, Phillips BA, Bo K, Galea MP. Physiotherapy as an adjunct to prolapse surgery: an assessor-blinded randomized controlled trial. Neurourol Urodyn. 2010 Jun;29(5):719-25. doi: 10.1002/nau.20828. PMID 19816918